CLINICAL TRIAL: NCT03901911
Title: Prevalence of Periodontitis on a Sample of Adult Egyptian Population: A Cross-sectional Study I
Brief Title: Prevalence of Periodontitis on a Sample of Adult Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Hamed Nada, B.Sc. in Oral and Dental Medicine, Cairo University
Other Study IDs: CEBD-CU-2018-12-13
Record Dates: First submitted 2019-01-20; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational cross-sectional study

DETAILED DESCRIPTION:
Adult patients will be included by consecutive manner from the diagnostic center at the Faculty of Dentistry.

All the patient information and medical history will be obtained from the patient and recorded byte principal investigator of this study.

Dental examinationof permanent fully erupted teeth will be performed by the principal investigator of this study, excluding third molars, retained roots, and implants.

Periodontal examinations will be performed using full-mouth periodontal examination (FMEP) methodology.

Periodontitis is defined here as 1-2 mm clinical attachment loss (CAL)in interproximal area in two non-adjacent teeth and Staging involves four categories (stages 1 through 4) and is determined after considering several variables including clinical attachment loss, amount and percentage of bone loss, probing depth, presence and extent of angular bony defects and furcation involvement, tooth mobility, and tooth loss due to periodontitis.

Grading includes three levels (grade A - low risk, grade B - moderate risk, grade C - high risk for progression) and encompasses, in addition to aspects related to periodontitis progression, general health status, and other exposures such as smoking or level of metabolic control in diabetes.

Aim of the Study will be explained to the patient, and informed consent will be given to him to sign and will be maintained with the rest of the data .

The evaluated parameters will be: clinical attachment loss (CAL), probing depth (PD), bleeding on probing (BOP), gingival recession (GR), plaque index (PI), furcation involvement ,tooth mobility and radiographic examination.

(CAL)will be Measured from the CEJ to the bottom of the gingival sulcus using Williams marking probe.

PD will be measured at six sites per tooth (mesiobuccal,mid-buccal, distobuccal, mesiolingual, mid-lingual and distolingual), PD will be measured as the distance from the cemento enamel junction (CEJ) to the bottom of the pocket using Williams marking probe.

GR will be measured as the distance from the CEJ to the free gingival margin, and this assessment will be assigned negative sign if the gingival margin is located coronally to the CEJ using Williams marking probe.

BOP gentle probing of the orifice of the gingival crevice. The periodontal probe will be inserted 1 to2 mm into the gingival sulcus starting at one interproximal area and moving to the other. If bleeding occurs within 10 seconds a positive finding is recorded.

PI the measurement of the state of oral hygiene by Silness-Löe Plaque index is based on recording both soft debris and mineralized deposits on the teeth using Williams marking probe. Missing teeth are not substituted.

0 No plaque

1 A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.

2 Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eye.

3 Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

Furcation involvement will be measured according to Glickman,1953 using Naber's Furcation Probe.

Radiographic examination will be performed by periapical radiograph for the most affected area to measure the linear measurement of bone loss & calculate the percentage of bone loss.

According to the Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions :

In grade A, there is slow rate of progression where the percentage of bone loss divided by age is less than 0.25.

In grade B there is a moderate rate of progression where the percentage of bone loss divided by age is from 0.25 to 1.0.

In grade C there is a rapid rate of progression where the percentage of bone loss divided by age is greater than 1.0.

ELIGIBILITY:
Inclusion Criteria:

• All Adult patients attending at the diagnostic center at the Faculty of Dentistry above 18 years old.

Exclusion Criteria:

* patients undergone periodontal therapy in the last 6 months.
* patients with psychomotor dysfunction.
* Patients less than 18 years old.
* Edentulous patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients attending at the diagnostic center at the Faculty of Dentistry above 18 years old.
Sampling Method: Probability Sample
Enrollment: 1708 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of periodontitis in percentage | 6 MONTHS
  Prevalence of periodontitis on a Sample of Adult Egyptian Population through determining clinical attachment loss.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490